CLINICAL TRIAL: NCT00719212
Title: A Multicenter Open Label Phase II Study of the Efficacy and Safety of AMG 479, a Fully Human Monoclonal Antibody Against Insulin-like Growth Factor Type 1 Receptor (IGF-1R) as Second Line Therapy in Patients With Recurrent Platinum Sensitive Ovarian Cancer
Brief Title: Study of AMG 479 as Second Line Therapy in Patients With Recurrent Platinum-sensitive Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research in Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIO 015
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Results first posted 2015-12-01 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — ganitumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMG 479 (Experimental): AMG 479 administered on day 1 of each 21-day cycle up to disease progression, unacceptable toxicity, withdrawal of consent or sponsor decision to stop the study.
  Interventions: Biological: AMG 479

INTERVENTIONS:
Biological: AMG 479 — Solution for infusion - 18 mg/kg on day 1 of each 21-day cycle

SUMMARY:
The purpose of this study is to obtain an estimate of the objective response rate (ORR) of AMG 479 in patients with recurrent platinum-sensitive ovarian epithelial (including fallopian tube and primary peritoneal) carcinoma failing frontline chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed ovarian epithelial (including fallopian tube and primary peritoneal) carcinoma. Baseline paraffin embedded tissue from the patient's primary diagnosis is requested before study enrollment and should be forwarded to the designated central laboratory. In patients with measurable disease or sufficient ascites, fresh frozen tissue or ascites fluid should be obtained by needle biopsy and submitted to the designated central laboratory.
* Prior treatment with at most 1 treatment regimen in the primary treatment setting.
* Platinum-sensitive disease defined by recurrence or progression of disease > 6 months AND < 24 months after completion of prior platinum based chemotherapy.
* Female > 18 years of age or legal age.
* ECOG performance status ≤ 1.
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Subjects with non-measurable disease with a biochemical recurrence are eligible provided the CA 125 is elevated by more than 2 times the upper limits of normal, confirmed in two successive samples, drawn at least one week apart.
* Resolution of any toxic effects of prior therapy (except alopecia) to NCI CTCAE v.3.0 Grade ≤ 1 and to baseline laboratory values as defined in the inclusion criterion immediately below.
* Adequate organ and bone marrow function
* Nondiabetic patients or Type 1 or 2 Diabetic Patients controlled with HgbA1c < 8% and fasting blood glucose level <160 mg/dL
* Adequate coagulation parameters (within 21 days prior to registration), International Normalized Ratio (INR) ≤1.5; Activated ProThrombin Time (APTT) ≤ 1.5 x ULN.

Exclusion Criteria:

* More than 1 prior chemotherapy regimen in the treatment of ovarian cancer.
* Platinum-resistant disease as defined by a recurrence or progression less or equal to six months after completion of the frontline platinum based chemotherapy.
* Anticipation of a need for a major surgical procedure (e.g., impending bowel obstruction, gastrointestinal perforation) or radiation therapy during the trial.
* Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or for in situ carcinoma of the cervix uteri.
* Prior treatment with investigational treatment targeted to IGF axis including, but not limited to, CP 751,871, IM-A12, RO4858696.
* Previous exposure to AMG 479.
* History of hypersensitivity to recombinant proteins.
* Prior treatment with a humanized monoclonal antibody.
* Treatment with chemotherapy, radiotherapy, surgery, blood products, or an investigational agent within 3 weeks of trial enrolment.
* Any of the following within 6 months prior to trial registration: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, NYHA class III or IV congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or other thromboembolic event.
* History of brain metastases, spinal cord compression, or carcinomatous meningitis.
* Patient of child-bearing potential is evidently pregnant (eg, positive human chorionic gonadotropin test) or is breast feeding.
* Patient of child-bearing potential is not willing to use adequate contraceptive precautions.
* Known active infection, or on antiretroviral therapy for HIV disease.
* Known positive test for chronic hepatitis B or C infection.
* Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the trial.
* Refusal or inability to give informed consent to participate in the trial.
* Other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the patient's safety, inhibit protocol participation, or interfere with interpretation of trial results, and in the judgment of the investigator would make the patient inappropriate for entry into this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gottfried E Konecny, MD, Study Chair — University of California, Los Angeles
Locations (37):
- United States (16):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - St Jude Heritage Healthcare, Fullerton, California
  - Wilshire Oncology Medical Group Inc, La Verne, California
  - LAC/USC Medical Center, Los Angeles, California
  - University of Southern California/ Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - North Valley Hematology/ Oncology Medical Group, Northridge, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Central Hematology Oncology Medical Group Inc., Pasadena, California
  - University of Colorado, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - St Joseph Mercy Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Comprehensive Cancer Centre of Nevada, Henderson, Nevada
- Canada (4):
  - Tom Baker Centre, Calgary
  - Juravinski Cancer Center, Hamilton
  - CHUM Hôpital Notre Dama, Montreal
  - Jewish General Hospital, Montreal
- France (5):
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - Centre Léon Berard, Lyon
  - Clinique Hartmann, Neuilly-sur-Seine
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Charité Campus Benjamin Franklin, Berlin
  - Universitatsklinikum Erlangen, Erlangen
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
- Ireland (5):
  - Cork University Hospital, Cork
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital, Dublin
  - St Jame's Hospital, Dublin
  - Waterford Regional Hospital, Waterford
- Kaplan Medical Center, Rehovot, Israel
- Spain (3):
  - Hospital Universitario de Tenerife, La Laguna (Santa Cruz de Tenerife)
  - Hospital U 12 de Octubre, Madrid
  - Hospital Universitario Virgen Macarena de Sevilla, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted over a total of 35 sites in 7 countries.
Period: Overall Study
Arm/Group | AMG 479
Started | 61
Completed | 17
Not Completed | 44
Not completed — Death | 41
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | AMG 479
Number analyzed (Participants) | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
  Canada | 7
  Germany | 4
  France | 24
  Ireland | 7
  Israel | 1
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Number; unit: participants] — 6-point (0 to 5) ordinal scale to assess how the disease affects the daily living abilities of the patient and determine apporpriate treatment and prognosis
  participants
    PS 0 (fully active) | 41
    PS 1 (restricted in physically strenuous activity) | 20
Time from initial diagnosis to registration [Mean (Standard Deviation); unit: Months] | 20.4 (6.2)
Origin of tumor [Number; unit: participants]
  Primary Peritoneal | 5
  Fallopian Tube | 3
  Ovarian | 46
  Ovarian + Primary Peritoneal | 3
  Ovarian + Fallopian Tube | 4
Stage at First Diagnosis (International Federation of Gynecology and Obstetrics (FIGO) ) [Number; unit: participants] — 5-point ordinal scale to assess the extent of the disease (0 ->IV). Roman numeral staging from the less to the most advanced cancer. Individual stage (I to III) is broken down in substage: IA, IB, IC,...
  participants
    IC | 3
    IIA | 1
    IIB | 2
    IIC | 2
    IIIA | 1
    IIIB | 3
    IIIC | 44
    IV | 5
Histopathologic Type [Number; unit: participants]
  Papillary serous | 42
  Mucinous | 2
  Endometroid | 5
  Clear cell | 4
  Mixed | 2
  Other | 6
Histologic Grade (G) [Number; unit: participants] — Cancer cells compared with normal cells
  participants
    G1 (well differentiated) | 1
    G2 (moderately differentiated) | 6
    G3 (poorly differentiated) | 45
    Not done | 9
CA 125 status [Number; unit: participants] — CA 125 level measurement from a blood sample
  participants
    With elevated CA 125 only | 5
    With elevated CA 125 + Non target lesion(s) only | 11
    With elevatCA125+target lesions+/-nontargetlesions | 37
    With CA125normal+target lesions+/-nontargetlesions | 8
Number of prior therapies [Number; unit: participants] — Prior anti-tumor treatment characteristics
  participants
    1 therapy | 2
    2 therapies | 38
    3 therapies | 16
    4 therapies | 3
    5 therapies | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Investigator Assessment: % of Patients in the Group Who Achieve a Complete Response(CR) or Partial Response(PR) According to RECIST Criteria and GCIG CA125 Response Criteria. - Assessments of the Response by the Investigators
Description: RECIST(v1.0):CR:disappearance of all target lesions or disappearance of all nontarget lesions & normalization of tumor marker level/•PR:at least 30% decrease in the sum of the longest diam(LD) of target les° taking as ref the baseline sum LD OR CR for target les° & incomplete response/SD for nontarget les°.
  CR & PR to be confirmed no less than 4 wks after initial doc of response.The def of the resp acc to serum CA125 level was as per GCIGCA125 criteria:
  * PR:elevated CA125 at baseline PR considered if a ≥ 50% decrease compared to baseline value was observed on 2 consecutive assessmts drawn at least 1 wk apart
  * CR:elevated CA125 at baseline CR was def with 2 CA125 values below ULN observed on 2 consecutive assessmts drawn at least 1 wk apart A pt was considered to have a best overall resp of:CR:if CR as per RECIST & CA125 /-PR: if CR as per RECIST & PR as per CA125 OR CR as per RECIST and SD as per CA125 with elevated CA125 at baseline OR PR as per RECIST & CR/PR or SD as per CA125
Time Frame: Radiological Tumor assessment: Every 9 (+/- 1 ) weeks during study treatment until documentation of progression or end of study treatment + confirmation PR or CR no less than 4 weeks after initial documentation of response + CA 125: Day 1 of each cycle
Population: Intent To Treat
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | AMG 479
Number analyzed (Participants) | 61
percentage of patients | 1.6 [0.0 to 8.8]

2. Secondary Outcome: Time To Progression (TTP) Investigator Assessment
Description: Interval from the date of registration to the date of disease progression Investigator assessment As per RECIST (v1.0), disease progression represented an increase of at least 20% in the sum of the longest diameter (SLD) of target lesions, taking as reference the smallest SLD recorded since the treatment started or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Every 9 (+/- 1 ) weeks during study treatment until documentation of progression or end of study treatment + confirmation PR or CR no less than 4 weeks after initial documentation of response
Population: Intent To Treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AMG 479
Number analyzed (Participants) | 61
months | 2.037 [1.906 to 2.168]

3. Primary Outcome: Objective Response Rate (ORR) Independent Radiology Committee % of Patients in the Group Who Achieve a Complete or Partial Response According to RECIST Criteria and GCIG CA 125 Response Criteria.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Intent To Treat
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | AMG 479
Number analyzed (Participants) | 61
percentage of patients | 1.6 [0.0 to 8.8]

4. Secondary Outcome: Clinical Benefit Rate (CBR) Investigator Assessmt % of Patients in the gp Who Achieve a Complete Response-CR,Partial Response-PR or Stable Disease-SD for 16wks From Registrat° Considering the Global Response Combining RECIST Criteria and CA125 Assessmts
Description: RECIST(v1.0):
  * CR:disappearance of all target les°&non-target les°&normalization of tumor marker level
  * PR:at least 30% decrease in the sum of the LD of target les°-ref the baseline sum LD OR CR for target les°&incomplete resp/SD for non target les°
  * SD:insufficient shrinkage for PR or increase for PD-ref the smallest sum LD since ttmt started or Persistence of one/more non-target les°or/&maintenance of tumor marker level above the normal
  CA125 level:
  * PR:elev of CA125 at baseline PR if a ≥ 50% decrease compared to baseline value observed on 2 consec assessmts drawn at least 1 wk apart
  * CR:elev of CA125 at baseline CR 2 CA125 below ULN observed on 2 consec assessmts drawn at least 1 wk apart
  * SD:neither CR/PR nor PD
  Best overall resp of :
  * CR:if CR per RECIST & per CA125
  * PR:if CR per RECIST & PR per CA125 OR CR per RECIST and SD per CA125 with elev CA125 at baseline OR PR per RECIST & CR/PR or SD per CA125
  * SD:other cases not qualifying for progression-at least 24 wks
Time Frame: At 16 weeks from registration
Population: Intent To Treat
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | AMG 479
Number analyzed (Participants) | 61
percentage of patients | 1.7 [0.0 to 8.9]

5. Secondary Outcome: Overall Survival (OS) Investigator Assessment
Description: Interval between the date of registration and the date of death
Time Frame: Day 1 of each cycle during study treatment + follow-up every 6 months for the first 3 years in the study or until death whichever occurs first
Population: Intent To Treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AMG 479
Number analyzed (Participants) | 61
months | 20.994 [19.450 to NA] — The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.

6. Secondary Outcome: Time To Marker Progression (TTMP) Investigator Assessment - Interval Form the Date of Registration to the Date of Disease Progression as Per GCIG 2005 Definition of CA 125 Progression.
Description: The GCIG criteria (November 2005) were used to define progressive disease, based on serum CA 125 levels, as follows:
  * Patients with elevated CA 125 pretreatment and normalization of CA 125 needed to show evidence of CA 125 greater than, or equal to, two times the ULN on two occasions at least 1 week apart or
  * Patients with elevated CA 125 pretreatment, which never normalizes needed to show evidence of CA 125 greater than, or equal to, two times the nadir value on two occasions at least 1 week apart or
  * Patients with CA 125 in the normal range pretreatment needed to show evidence of CA 125 greater than, or equal to, two times the ULN on two occasions at least 1 week apart.
Time Frame: Day 1 of each cycle
Population: Intent To Treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AMG 479
Number analyzed (Participants) | 61
months | 4.961 [2.760 to 12.813]

7. Secondary Outcome: Progression-free Survival (PFS) Investigator Assessment - Interval From Registration to Disease Progression or Death Due to Any Cause - According to RECIST and CA 125
Description: A patient may have been declared to have progressive disease on the basis of radiological measuremt of tumor lesions assessmt or CA125 evaluation (tumor measuremts taking precedence).Radiological progression was defined as per the RECIST guidelines (Therasse et al, JNCI2000) as at least 20% increase in the sum of the longest diameters of target lesions(ref the smallest sum of the longest diam recorded since the treatmt started or since the appearance of at least 1 new lesion).Serum CA125 progression was defined, according to the 2005 GCIG def: pts with:
  * Elevated CA125 pretreatmt and normalization of CA125 has to show evidence of CA125≥ 2 times the upper normal limit on 2 occasions at least 1 wk apart OR
  * Elevated CA125 pretreatmt which never normalized must show evidence of CA125≥ 2 times the nadir value on 2 occasions at least 1 wk apart OR
  * CA125 in the normal range pretreatmt had to show evidence of CA125 ≥ 2 times the upper normal limit on 2 occasions at least 1 wk apart
Time Frame: as for outcome 2
Population: Intent To Treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AMG 479
Number analyzed (Participants) | 61
months | 1.938 [1.446 to 2.103]

ADVERSE EVENTS:
Arm/Group | AMG 479
Serious Adverse Events (participants affected / at risk) | 12/61
Other Adverse Events (participants affected / at risk) | 60/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMG 479 (N=61)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Candida Infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMG 479 (N=61)
Abdominal distension (Gastrointestinal disorders) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 19 (24)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 15 (16)
Diarrhoea (Gastrointestinal disorders) | 17 (24)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 8 (10)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 16 (27)
Stomatitis (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 9 (13)
Asthenia (General disorders) | 15 (19)
Chest pain (General disorders) | 4 (7)
Chills (General disorders) | 8 (12)
Fatigue (General disorders) | 21 (25)
Pyrexia (General disorders) | 5 (6)
Hypersensitivity (Immune system disorders) | 8 (9)
Urinary tract infection (Infections and infestations) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Dizziness (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 10 (14)
Anxiety (Psychiatric disorders) | 4 (5)
Depression (Psychiatric disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No